CLINICAL TRIAL: NCT05269381
Title: A Phase I/II Study of Personalized Neoantigen Peptide-Based Vaccine in Combination With Pembrolizumab in Advanced Solid Tumors (PNeoVCA)
Brief Title: Personalized Neoantigen Peptide-Based Vaccine in Combination With Pembrolizumab for Treatment of Advanced Solid Tumors
Acronym: PNeoVCA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210102; NCI-2022-01258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-008509 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Merkel Cell Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Merkel Cell Carcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Locally Advanced Cervical Carcinoma; Locally Advanced Endometrial Carcinoma; Locally Advanced Gastric Adenocarcinoma; Locally Advanced Gastroesophageal Junction Adenocarcinoma; Locally Advanced Head and Neck Squamous Cell Carcinoma; Locally Advanced Hepatocellular Carcinoma; Locally Advanced Lung Non-Small Cell Carcinoma; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Melanoma; Locally Advanced Merkel Cell Carcinoma; Locally Advanced Renal Cell Carcinoma; Locally Advanced Skin Squamous Cell Carcinoma; Locally Advanced Triple-Negative Breast Carcinoma; Locally Advanced Unresectable Breast Carcinoma; Locally Advanced Unresectable Cervical Carcinoma; Locally Advanced Unresectable Gastric Adenocarcinoma; Locally Advanced Unresectable Gastroesophageal Junction Adenocarcinoma; Locally Advanced Unresectable Renal Cell Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Cervical Carcinoma; Metastatic Endometrial Carcinoma; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hepatocellular Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Merkel Cell Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Skin Squamous Cell Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Metastatic Urothelial Carcinoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Merkel Cell Carcinoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IV Merkel Cell Carcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Skin Squamous Cell Carcinoma; Stage III Cervical Cancer AJCC v8; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Hepatocellular Carcinoma AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8; Triple-Negative Breast Carcinoma; Unresectable Cervical Carcinoma; Unresectable Endometrial Carcinoma; Unresectable Gastric Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma; Unresectable Head and Neck Squamous Cell Carcinoma; Unresectable Hepatocellular Carcinoma; Unresectable Lung Non-Small Cell Carcinoma; Unresectable Malignant Solid Neoplasm; Unresectable Melanoma; Unresectable Merkel Cell Carcinoma; Unresectable Renal Cell Carcinoma; Unresectable Skin Squamous Cell Carcinoma; Unresectable Triple-Negative Breast Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Lung Neoplasms | interventions — Cyclophosphamide; pembrolizumab; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, vaccine, pembrolizumab) (Experimental): Patients receive cyclophosphamide IV on day -3. Patients then receive personalized neoantigen vaccine with sargramostim SC on days 1, 4, 8, and 15 of cycle 1 and day 1 of cycles thereafter. Patients also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients may undergo blood sample collection during screening, cycle 1 days -3, 1, 8, 15, 22, cycles 2, 3, 4, 5, 7, 8 and 9+ day 1 and 30 days after last dose of GM-CSF or pembrolizumab and may undergo tissue biopsy during screening, week 25 or at the time of disease progression. Patients also undergo CT or MRI during screening, week 9 then every 9 weeks, and 30 days after last dose of GM-CSF or pembrolizumab.
  Interventions: Drug: Cyclophosphamide; Biological: Neoantigen Peptide Vaccine; Biological: Pembrolizumab; Biological: Sargramostim

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Neoantigen Peptide Vaccine — Receive personalized neoantigen vaccine SC
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial tests the safety and tolerability of an experimental personalized vaccine when given by itself and with pembrolizumab in treating patients with solid tumor cancers that have spread to other places in the body (advanced). The experimental vaccine is designed target certain proteins (neoantigens) on individuals' tumor cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving the personalized neoantigen peptide-based vaccine with pembrolizumab may be safe and effective in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of personalized neoantigen peptide vaccine in combination with pembrolizumab in advanced solid cancers.

SECONDARY OBJECTIVES:

I. To evaluate the feasibility of personalized neoantigen peptide vaccine in combination with pembrolizumab in advanced solid cancers.

II. To obtain preliminary information on the immunogenicity of neoantigen in induction of specific cellular immune responses and humoral immune response.

EXPLORATORY OBJECTIVES:

I. To obtain preliminary estimates of efficacy as measured by objective response rate (ORR based on Response Evaluation Criteria in Solid Tumors [RECIST]) of personalized neoantigen peptide vaccine and pembrolizumab in patients with selected advanced solid tumors.

II. To obtain preliminary information of immunity persistence, as well as pre-existing immunity.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) on day -3. Patients then receive personalized neoantigen vaccine with sargramostim (GM-CSF) SC on days 1, 4, 8, and 15 of cycle 1, and day 1 of cycles thereafter. Patients also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months up to 2 years from study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION COHORT 1 ONLY: Histologically confirmed unresectable locally advanced or metastatic solid malignancies
* PRE-REGISTRATION COHORT 1 ONLY: Has cancer progression after at least one line of standard of care systemic treatment
* PRE-REGISTRATION COHORT 2 ONLY: Histologically confirmed unresectable locally advanced or metastatic solid malignancies that pembrolizumab is Food and Drug Administration (FDA) approved indication including melanoma, non-small cell lung cancer (NSCLC), head and neck squamous cell cancer (HSNCC), urothelial carcinoma, any microsatellite instability (MSI)-high tumor, gastric or gastroesophageal junction (GEJ) adenocarcinoma, cervical cancer, hepatocellular carcinoma (HCC), merkel cell carcinoma (MCC), renal cell carcinoma (RCC), endometrial carcinoma, tumor mutational burden-high (TMB-H) cancer, cutaneous squamous cell carcinoma (cSCC), and triple-negative breast cancer (TNBC) or other solid tumors that will benefit from pembrolizumab per the treating physician's judgment.
* PRE-REGISTRATION COHORT 2 ONLY: Patient is eligible to receive pembrolizumab with or without chemotherapy per the treating physician's judgement or has been on pembrolizumab through compassionate use
* PRE-REGISTRATION: Age >= 18 years
* PRE-REGISTRATION: Willing to provide mandatory tissue specimens per protocol

  * NOTE: This includes mandatory fresh tissue specimen at pre-registration for complete exome and transcriptome sequencing unless patient had sequencing under Mayo Institutional Review Board (IRB) protocol #13-000942, #14-004094, or #21-007742 and has been identified for potential production of REAL Neo vaccine. Patients who had sequencing under Mayo IRB protocol #13-000942, #14-004094, or #21-007742 and have been identified for potential production of REAL Neo vaccine are allowed to proceed with neoantigen production.
* PRE-REGISTRATION: Measurable disease as defined by RECIST (version 1.1) criteria

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease or non-measurable disease
* PRE-REGISTRATION: Patients with actionable genomic abnormality including, but not limited to EGFR, ALK, MET, ROS-1, RET, NTRK, KRAS or BRAF must have also received and progressed on at least one line of prior FDA-approved targeted therapy
* PRE-REGISTRATION: Provide written informed consent
* PRE-REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* PRE-REGISTRATION: Willing to provide mandatory blood specimens for correlative research
* PRE-REGISTRATION: Negative pregnancy test done =< 7 days prior to pre-registration for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* PRE-REGISTRATION: Willing to employ a highly effective method of contraception from the time of pre-registration through 6 months after the final vaccine cycle
* PRE-REGISTRATION: Willing to receive a tetanus vaccination if subject has not had one =< 1 year prior to pre-registration
* PRE-REGISTRATION: Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* PRE-REGISTRATION: Anticipated life expectancy of > 6 months
* PRE-REGISTRATION: Recovered from all toxicities associated with prior treatment to acceptable baseline status (for laboratory toxicity see below limits for inclusion) or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, Grade of 0 or 1, except for toxicities not considered a safety risk per treating investigator (e.g., alopecia or vitiligo).
* PRE-REGISTRATION: Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to pre-registration) (Must be >= 7 days after most recent transfusion)
* PRE-REGISTRATION: Absolute neutrophil count (ANC) >= 1500/mm^3 or >= 1.5 X 10^9/L (obtained =< 28 days prior to pre-registration)
* PRE-REGISTRATION: Platelet count >= 100,000/mm^3 or >= 100 X 10^9/L (obtained =< 28 days prior to pre-registration) (Must be >=7 days after most recent transfusion)
* PRE-REGISTRATION: Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 28 days prior to pre-registration)
* PRE-REGISTRATION: Aspartate transaminase (AST) and alanine transaminase (ALT) =< 3 x ULN or =< 5 x ULN for patients with liver metastases (obtained =< 28 days prior to pre-registration)
* PRE-REGISTRATION: Creatinine =< 1.5 x ULN OR calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 28 days prior to pre-registration)
* PRE-REGISTRATION: International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy in which case PT or PTT must be within target range of therapy (obtained =< 28 days prior to pre-registration)
* REGISTRATION COHORT 1 ONLY: Histologically confirmed unresectable locally advanced or metastatic solid malignancies
* REGISTRATION COHORT 1 ONLY: Has cancer progression after at least one line of standard of care systemic treatment
* REGISTRATION COHORT 2 ONLY: Histologically confirmed unresectable locally advanced or metastatic solid malignancies that pembrolizumab is FDA approved indication (including melanoma, non-small cell lung cancer (NSCLC), head and neck squamous cell cancer (HSNCC), urothelial carcinoma, any microsatellite instability (MSI)-high tumor, gastric or gastroesophageal junction (GEJ) adenocarcinoma, cervical cancer, hepatocellular carcinoma (HCC), merkel cell carcinoma (MCC), renal cell carcinoma (RCC), endometrial carcinoma, tumor mutational burden-high (TMB-H) cancer, cutaneous squamous cell carcinoma (cSCC), and triple-negative breast cancer (TNBC) or other solid tumors that will benefit from pembrolizumab per the treating physician's judgement.
* REGISTRATION COHORT 2 ONLY: Pembrolizumab without chemotherapy remains as a reasonable treatment option at the treating physician's decision
* REGISTRATION: Age >= 18 years
* REGISTRATION: Soft tissue lesion amenable for adequate tissue sampling

  * NOTE: It should not be tumor which was radiated in the past.
* REGISTRATION: Successful sequencing and production of REAL-Neo vaccine
* REGISTRATION: Measurable disease as defined by RECIST (version 1.1) criteria

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease or non-measurable disease
* REGISTRATION: ECOG Performance Status (PS) 0 or 1
* REGISTRATION: Anticipated life expectancy of > 6 months
* REGISTRATION: Hemoglobin >= 9.0 g/dl (obtained =< 14 days prior to registration)
* REGISTRATION: Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* REGISTRATION: Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* REGISTRATION: Total bilirubin =< 1.5 x ULN (obtained =< 14 days prior to registration)
* REGISTRATION: Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* REGISTRATION: PT/INR and aPTT =< 1.5 x ULN unless patient is receiving anticoagulant therapy in which case INR or aPTT must be within target range of therapy (obtained =< 14 days prior to registration)
* REGISTRATION: Calculated creatinine clearance >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* REGISTRATION: Provide written informed consent
* REGISTRATION: Willing to provide mandatory blood specimens for correlative research
* REGISTRATION: Willing to provide mandatory tissue specimens for correlative research
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* REGISTRATION: Patients with actionable genomic abnormality including, but not limited to EGFR, ALK, MET, ROS-1, RET, NTRK, KRAS or BRAF must have also received and progressed on at least one line of prior FDA-approved targeted therapy
* REGISTRATION: Negative pregnancy test done =< 14 days prior to registration for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* REGISTRATION: Willing to employ a highly effective method of contraception from the time of pre-registration through 6 months after the final vaccine cycle
* REGISTRATION: Willing to receive a tetanus vaccination if subject has not had one =< 1 year prior to pre-registration
* REGISTRATION: Recovered from all toxicities associated with prior treatment to acceptable baseline status (for laboratory toxicity see below limits for inclusion) or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0, Grade of 0 or 1, except for toxicities not considered a safety risk per treating investigator (e.g., alopecia or vitiligo)

Exclusion Criteria:

* PRE-REGISTRATION: Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant person
  * Nursing person unwilling to stop breast feeding
  * Person of childbearing potential who are unwilling to employ adequate contraception from the time of registration through 6 months after the final vaccine cycle
* PRE-REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* PRE-REGISTRATION: History of myocardial infarction =< 6 months prior to pre-registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
* PRE-REGISTRATION: Acute, reversible effect(s) of prior therapy not recovered to baseline regardless of interval since last treatment
* PRE-REGISTRATION: Uncontrolled illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Congestive heart failure with New York Heart Association class III or IV; moderate to severe objective evidence of cardiovascular disease
  * Stroke =< 3 months prior to pre-registration
  * Significant cardiac arrhythmia or unstable angina
  * Any other conditions that would limit compliance with study requirements
* PRE-REGISTRATION: Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* PRE-REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm, except for pembrolizumab
* PRE-REGISTRATION: Any prior hypersensitivity or adverse reaction to GM-CSF
* PRE-REGISTRATION: Other active malignancy =< 3 years prior to pre-registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* PRE-REGISTRATION: Known history of active autoimmune disease that has required systemic treatment in the =<30 days (i.e., with use of disease modifying agents, corticosteroids >10 mg daily prednisone equivalent, or other immunosuppressive drugs) prior to pre-registration.

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with celiac disease controlled with diet modification are not excluded
* REGISTRATION: Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* REGISTRATION: Any of the following prior therapies:

  * Chemotherapy, experimental drugs (except for pembrolizumab), or small molecules inhibitors (except for endocrine therapies) =< 3 weeks prior to registration
  * Radiation =< 2 weeks prior to registration
  * Major Surgery =< 4 weeks prior to registration
  * Received a live vaccine =< 30 days prior to registration
  * NOTE: Recent anti-PD1 or anti-PD-L1, such as pembrolizumab, nivolumab, atezolizumab, and durvalumab, is allowed, but the last dose of anti-PD-1 or anti-PD-L1 treatment should be more than 21 days from first dose of vaccination on the study (for Cohort 2 only)
  * Palliative radiation therapy for symptoms control including, but not limited to, bone metastatic lesion radiation therapy is allowed, but the last dose of radiation therapy should be more than 14 days from the first dose of vaccination on the study
* REGISTRATION: CTCAE >= Grade 3 treatment-emergent adverse event (TEAE) to prior checkpoint inhibitor, TEAE requiring systemic corticosteroids (> 10 mg daily prednisone equivalent), or permanent treatment discontinuation due to toxicity
* REGISTRATION: Neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy), or a history of rhabdomyolysis
* REGISTRATION: Active autoimmune diseases that require chronic systemic steroids (> 10 mg daily prednisone equivalent) or immunosuppressive agents
* REGISTRATION: Requirement for systemic corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications =< 14 days prior to registration

  * NOTE: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* REGISTRATION: Evidence of leptomeningeal disease
* REGISTRATION: Central nervous system metastases that are untreated, symptomatic, or require steroids > 10 mg daily prednisone equivalent

  * NOTE: Patients with history of stable treated brain metastases are eligible. Stable treated metastases are defined as follows: No evidence of progression for >= 4 weeks on brain imaging (either magnetic resonance imaging [MRI] or computed tomography [CT] scan)
* REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years from first vaccine administration
  The maximum grade for each type of adverse event will be recorded for each patient. The attribution, grade, and type of adverse event (AE), the dose level, the tumor type, and the prior treatment will be tabulated for each patient

SECONDARY OUTCOMES:
The number and percentage of participants who completed the sequencing with satisfactory data quality registration and identified at least 10 actionable peptides, meet the eligibility criteria for registration, and able to initiate vaccine production | Up to 16 weeks
  Feasibility will be defined as the number and percentage of participants who completed the sequencing with satisfactory data quality registration and identified at least 10 actionable peptides, meet the eligibility criteria for registration, and able to initiate vaccine production within 16 weeks.
Immunogenicity responders | Within 24 weeks
  The number and percentage of patients who are vaccine immunity responders will be calculated. The immunity responder for each patient is defined as >= 20% of neoantigens formulated into vaccine with at least 3-fold of value increase at any timepoint,

OTHER OUTCOMES:
Objective response rate (ORR) | Within 12 weeks
  The total ORR (partial response [PR]+complete response [CR] rate) at the recommend dose will be reported. For each patient at the recommend dose, CR or PR will be confirmed based on at least two consecutive evaluations with 6 weeks apart or at the next re-staging scans if it is determined as reasonable by the treating physician.
Immunity persistency | Within 24 weeks from baseline
  The number of patients with immunity persistency will be summarized. Persistency of immunity for each patient is detected as at least 3-folds of value increase of neoantigen from baseline at 12 months among neoantigens that had been detected with at least 3-folds of value increase within 24 weeks from baseline
Pre-existing Immunity | Within 24 weeks from baseline
  The number of patients with pre-existing immunity will be summarized. A patient will be considered to have pre-existing immunity at baseline if the mean antigen-specific T cell frequency is statistically higher (P < 0.05) from no antigen wells.

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Lou, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials